CLINICAL TRIAL: NCT04793854
Title: Sickle Cell Disease, Neurocognitive Disorders, Social Participation
Acronym: SOCIODREP
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Collaborators: Université des Antilles, LAboratoire ACTES (Unknown)
Responsible Party: Sponsor
Other Study IDs: PAP_RNI_2018/02
Record Dates: First submitted 2021-03-08; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Sickle Cell Disease
Keywords: neurocognitive disorders; social participation
MeSH Terms: conditions — Anemia, Sickle Cell; Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case: Children with sickle cell anemia attending the centre of reference for sickle cell disease in Guadeloupe.
  Interventions: Other: Measure of the Life habits (MHAVIE)
- Control: Control children without chronical disease
  Interventions: Other: Measure of the Life habits (MHAVIE)

INTERVENTIONS:
Other: Measure of the Life habits (MHAVIE) — Life habits include daily activities and social in 6 groups. Environmental factors include social (9 different subgroups) and physical factors (7 different subgroups).
  Personal factors are person related parameters (gender, age, sociocultural ethnic, skills, deficiencies factors,…).
  Other Names: Measure of Environmental Quality (MQE); semi-guided interviews

SUMMARY:
This project will promote the development of transdisciplinary analyses. Neuropsychological disorders will be explored with the usual appropriate tests done by psychologists and neuropsychologists regularly involved in the management of sickle cell disease affected children. For the social sciences' component, various methods will be used: Measure of the Life habits (MHAVIE), Measure of Environmental Quality (MQE) and semi-guided interviews will complete the collection of qualitative data. The expected results concern the identification of the barriers or facilitators the sickle cell patients might face in their social participation, whether they are affected or not by neurological disorders.

DETAILED DESCRIPTION:
Sickle cell anaemia, which is the most frequent genetic disease in France, requires an early and optimal care to reduce its morbidity and mortality. Children with sickle cell anaemia who are significantly anaemic may present neurological complications including stroke with or without clinical signs. A major risk associated to these strokes is the impairment of the general intellectual ability and learning ability, essentially resulting from neuropsychological disorders affecting intellectual functioning, executive and attentional functions. Although the negative impact of sickle cell anemia on the quality of life of the affected children and adolescents is well documented, no study has been focused on the role played by the neurocognitive disorders on their social participation. The objective of this project is the assessment of the influence of neurocognitive disorders in the social participation of children and adolescent with sickle cell anemia (6 to 16 years old), followed in Guadeloupe. This project will promote the development of transdisciplinary analyses. Neuropsychological disorders will be explored with the usual appropriate tests done by psychologists and neuropsychologists regularly involved in the management of sickle cell disease affected children. For the social sciences' component, various methods will be used: Measure of the Life habits (MHAVIE), Measure of Environmental Quality (MQE) and semi-guided interviews will complete the collection of qualitative data. The expected results concern the identification of the barriers or facilitators the sickle cell patients might face in their social participation, whether they are affected or not by neurological disorders

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell anemia
* Age between 6 and 16 years inccuded, attending the centre of reference for sickle cell disease in Guadeloupe
* Informed consent
* Medical insurance

Exclusion Criteria:

* Other sickle cell syndrome other than SS or Sb-thal
* Less than 6 years old or older than 16
* Attending other sickle cell departments
* No medical insurance

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: This study concerns patients with sickle cell anemia, followed by physicians in Guadeloupe.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2018-09-19 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
MHAVIE-Children | Inclusion
  Assessment of Life Habits-LIFE-H
MQE | Inclusion
  Measure of Environmental Quality (MQE)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de la Guadeloupe, Pointe-à-Pitre, France, Guadeloupe

IPD SHARING:
Plan to Share IPD: No